CLINICAL TRIAL: NCT04377750
Title: The Use of Tocilizumab in the Management of Patients Who Have Severe COVID-19 With Suspected Pulmonary Hyperinflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Sheba Medical Center (Other Government); Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0224-20-HMO-CTIL
Record Dates: First submitted 2020-04-23; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Covid19 Pneumonia
Keywords: SARS-CoV-2; Cytokine storm; IL-6
MeSH Terms: conditions — Cytokine Release Syndrome | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab treatment group (Experimental): Treatment: intravenous administration of monoclonal anti body anti- IL6R. The dose is 8 mg/kg up to total dose of 800 mg.
  Interventions: Drug: Tocilizumab
- Placebo group (Placebo Comparator): Placebo. intravenous administration of 100 ml of normal saline.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — The placebo treatment arm will include 100 ml of normal saline administered along 60 min
  Other Names: Placebo

SUMMARY:
Title: The use of Tocilizumab in the management of patients who have severe COVID-19 with suspected pulmonary hyperinflammation.

This is a study designed to assess the therapeutic value of intravenous tocilizumab administered as single 8mg/Kg dose in patients affected by SARS-CoV2 infection with a pulmonary manifestation causing hypoxia. Aim of the study is to test the hypothesis that anti-IL6 treatment can be effective in reducing the virus-induced cytokine storm, blocking deterioration of lung function or even promoting a rapid improvement of clinical conditions, preventing tracheal intubation and/or death.

This drug will be administered to those patients entering the ICU with severe acute respiratory failure COVID-19 disease. The endpoints are death and duration of hospitalization. The patients will be assessed with surrogate markers determining the level of the cytokine storm.

DETAILED DESCRIPTION:
Study design This is a multicenter, two arms, 2:1 (treatment: control) open-label randomized control study with a drug approved for another indication in Israel. All the patients enrolled will be treated with tocilizumab or not. One-month mortality rate is the primary endpoint. One arm will be the study drug anti-IL6R (Tocilizumab (Actmera)) 8 mg/kg given IV during one hour once. The placebo will be a 100 ml saline IV infusion administered along one hour.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender
2. Age 18 and older
3. Informed consent for participation in the study
4. Virological diagnosis of Sars-CoV2 infection (PCR)
5. Acute respiratory failure
6. Radiographic pneumonia, defined as any/ changing new lung infiltrate
7. Patient breathing spontaneously, required more than 50% oxygen and MEWS score > 7.
8. If intubated, intubated less than 24 hours with PaO2/Fio2 ratio ≤ 200 and PEEP ≥ 5 cm H2O.

Exclusion Criteria:

1. Known hypersensitivity to tocilizumab or its excipients
2. Patient with a life expectancy of less than 6 months.
3. Known active infections or other clinical condition that contra-indicate tocilizumab and cannot be treated or solved according to the judgement of the clinician.
4. Neutrophils <500 / mmc
5. Platelets <40.000 / mmc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
Survival | One-month
  One-month mortality rate .

CONTACTS AND LOCATIONS:
Overall Officials: Juli Benbenisty, MPH, Study Chair — Hadassah Medical Organization
Locations (4):
- Israel (4):
  - Hadassah Medical Orginisation, Jerusalem, Please Select:
  - Barzilai Medical Center, Ashkelon
  - Wolfson Medical Center, Holon
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No
No plan